CLINICAL TRIAL: NCT06415916
Title: Ultrasound and Clinical Approach for the Dynamic Assessment of Fluid Tolerance in the Intensive Care Unit : FLUID-REACT Study
Brief Title: Ultrasound and Clinical Approach for the Dynamic Assessment of Fluid Tolerance in the Intensive Care Unit
Acronym: FLUID-REACT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GUINOT 2024
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Volume Expander

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: Patients admitted to intensive care who require volume expander
  Interventions: Procedure: Cardiac ultrasound; Procedure: Lung ultrasound

INTERVENTIONS:
Procedure: Cardiac ultrasound — Performed 5 times between 0 and 120 minutes
Procedure: Lung ultrasound — Performed 5 times between 0 and 120 minutes

SUMMARY:
A major cause of admission to intensive care is acute circulatory failure resulting from organ hypoperfusion due to factors such as hypotension and myocardial dysfunction. The standard treatment, including volume expansion and vasopressor/inotropic agents, often leads to water and sodium overload, increasing the risk of morbidity and mortality in the ICU. The combination of this overload and myocardial dysfunction lead to venous congestion, particularly affecting the lungs, kidneys and gastrointestinal system. Effective fluid management is therefore crucial to maintain a balance between adequate tissue perfusion and prevention of fluid overload. Fluid tolerance, defined as a patient's ability to tolerate additional volumes of solutes without adverse effects, is assessed retrospectively by clinical signs (capillary refill time, oedema, hepatojugular reflux, etc.) and ultrasound scores (VExUS score, LUS score, etc.). However, these indicators do not fully reflect the complexity of venous congestion in patients with various conditions.

Assessing fluid tolerance remains a challenge in clinical practice. It requires a personalised approach and the use of dynamic tests such as passive leg raising to predict response to vascular filling. Despite their common use, there are no studies evaluating the ability of changes in congestion markers during passive leg raising to predict fluid tolerance.

In conclusion, the main hypothesis is that changes in ultrasound congestion parameters (VExUS score, LUS score and others) during passive leg raising could predict a patient's subsequent tolerance to volume expander.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who has provided non-opposition (or health proxy or a close relative if unable to receive the information)
* Patient admitted to intensive care and requiring volume expander

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant, parturient or breast-feeding women
* Poor echogenicity assessed by the operator
* Chronic AC/FA
* Mechanical cardiac assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified by the investigator on admission to the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
the variation in the VExUs score during passive leg raising | Through study completion, on average of 2 hours
  The VExUS score is calculated from ultrasound-doppler measurements of the inferior vena cava (IVC), suprahepatic venous flow (S wave, D wave), portal flow (continuous, pulsatile >30%, pulsatile >50%), renal venous flow (continuous, pulsatile biphasic, pulsatile monophasic). It is graded from 0 to 3

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France